CLINICAL TRIAL: NCT01523080
Title: An Open Label, Balanced, Randomised, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover Bioavailability Study Comparing Acetaminophen 650 mg Extended Release Gel Tabs (Containing Acetaminophen 650 mg) of OHM Laboratories Inc. (Subsidiary of Ranbaxy) With Tylenol 8 Hour Extended Release Gel Tabs (Containing Acetaminophen 650 mg) of McNeil Consumer & Speciality Pharmaceuticals in Healthy, Adult, Human, Male Subjects Under Fasting Condition
Brief Title: A Relative Bioavailability Study of Acetaminophen Extended Release Gel Tabs 650 mg Under Fasting Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Sponsor
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 104_ACETA_06
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tylenol® 650 mg (Active Comparator): Tylenol® 650 mg of McNeil Consumer and Specialty Pharmaceuticals, Division of McNeil PPC, INC. Fort Washington, PA 19034 USA.
  Interventions: Drug: Acetaminophen
- Acetaminophen extended release Gel tabs 650 mg (Experimental): Acetaminophen extended release Gel tabs 650 mg of OHM Laboratories Inc. (A subsidiary of Ranbaxy Pharmaceuticals Inc., USA)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Extended release Gel tabs 650 mg

SUMMARY:
The study was to compare single-dose oral bioavailability of acetaminophen 650 mg extended release geltabs (containing acetaminophen 650 mg) of OHM Laboratories Inc. (subsidiary of Ranbaxy Pharmaceuticals Inc., USA) with Tylenol 8 hour extended release gel tabs (containing acetaminophen 650 mg) of McNeil Consumer & Speciality Pharmaceuticals, U.S.A in healthy, adult, male human subjects under fasting condition.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single dose, crossover bioavailability study comparing acetaminophen 650 mg extended release gel tabs (containing acetaminophen 650 mg) of OHM Laboratories Inc. (subsidiary of Ranbaxy) with Tylenol 8 hour extended release gel tabs (containing acetaminophen 650 mg) of McNeil Consumer & Speciality Pharmaceuticals in healthy, adult, human, male subjects under fasting condition.

The treatments were assigned to the study subjects according to SAS generated randomization schedule. Each subject received a single oral dose either Test or Reference product in each period with 240ml of water at ambient temperature after an overnight fast of at least 10 hours under supervision of a trained study personnel.

During the course of the study, safety parameters inclusive of vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical, serology parameters and urine analysis) at base line were assessed. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.

Exclusion Criteria:

* History of hypersensitivity to Acetaminophen or to any of the components of the formulation.
* History of skin rashes, thrombocytopenia, urticaria or angioedema
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Presence of disease markers of HIV 1 or 2, Hepatitis B or C viruses or syphilis infection.
* Presence of values that were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates or cannabinoids)
* Presence of values, which were significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (> 4/HPF), epithelial cells (> 4/HPF), glucose (positive) or protein (positive).
* Clinically abnormal ECG or Chest X-ray.
* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma (rise of pressure inside the eye leading to blurring or loss of vision)
* History of any psychiatric illness, which might impair the ability to provide written informed consent.
* Regular smokers who smoked more than 10 cigarettes daily or had difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or had difficulty in abstaining for the duration of each study period.
* Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Participation in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 19 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax) of Acetaminophen | 0, 0.167, 0.33, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16 and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology Unit, Majeedia Hospital (2nd Floor), New Delhi, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html